CLINICAL TRIAL: NCT02780479
Title: Oral Dexamethasone Versus Oral Prednisone in Children Hospitalized With Asthma: A Randomized Control Study
Brief Title: Steroids in Children Hospitalized With Asthma
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: insufficient number of participants met the enrollment criteria.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UFJ 2016-24
Record Dates: First submitted 2016-05-19; First posted 2016-05-23 (Estimated); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Asthma; Status Asthmaticus; Wheezes
Keywords: Prednisone; Dexamethasone; Asthma exacerbation; Hospitalized
MeSH Terms: conditions — Asthma; Status Asthmaticus; Respiratory Sounds | interventions — Dexamethasone; Calcium Dobesilate; Prednisone; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone (Experimental): Dexamethasone arm: will receive second dose of oral Dexamethasone 0.6 mg/kg/dose max of 16 mg, 24 hour from the first dose given in emergency department.
  Interventions: Drug: Dexamethasone
- Prednisone (Active Comparator): Prednisone arm: will receive oral Prednisone 1mg/kg with max of 30 mg twice daily starting 24 hours after the Dexamethasone dose given in emergency department for 8 additional doses.
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Dexamethasone — at 24 hours from the first Dexamethasone dose given in ED.
  Other Names: Decadron
  Arms: Dexamethasone
Drug: Prednisone — at 24 hours from the first Dexamethasone dose given in ED.
  Other Names: Orapred
  Arms: Prednisone

SUMMARY:
Asthma is the most common chronic disease of children. A short (3-5 day) course of a short-acting steroid such as Prednisone or Prednisolone has long been the standard of care for asthma exacerbation. Dexamethasone efficacy in asthma exacerbation has been studied in the outpatient setting and was found to be as effective as Prednisone. Dexamethasone has the advantage of shorter course, more compliance, and more tolerable. This has led many emergency departments to provide a 1-2 dose course of Dexamethasone on discharge. Thus, many inpatients have received a first dose of Dexamethasone prior to reaching the inpatient unit, leading to confusion about the best plan for these patients. Many hospitalist pediatricians continue to give a 5-day total course with Prednisone, but some patients have begun to receive a second dose of Dexamethasone 24 hours after the first dose. To our knowledge, no studies have been done to compare the efficacy of these two protocols in pediatric patients requiring hospitalization. The hypothesis is that a second dose of Dexamethasone is as effective as four additional days of Prednisone in hospitalized children with asthma exacerbation. This is an open label, randomized control study comparing these treatments in children age 2-18 hospitalized with asthma exacerbation who have received a first dose of Dexamethasone.

DETAILED DESCRIPTION:
Corticosteroids are the first-line therapy for managing acute asthma exacerbations. Studies have shown that systemic steroids effect decrease relapse and hospital admission. Due to its short half-life, Prednisone is usually given daily or twice daily for 3-5 days. It has been associated with poor compliance due it the prolonged course. Dexamethasone half-life is 36 - 72 hours.

Several studies have shown no difference in outcomes between 3-5 days of prednisone and different forms of dexamethasone, including single intramuscular dose or single oral dose or two oral doses 1 day apart. However, those studies were done in the emergency department (ED). Lack of response to initial asthma treatment in ED results in admission to the hospital, implying more severe exacerbation than those able to be discharged. Some clinician shift to oral prednisone once admitted to the floor for patients who have received Dexamethasone or not. Others have begin to complete the Dexamethasone course with one more dose of Dexamethasone 24 hour after the first dose. Dexamethasone has the advantage of compliance and tolerability, however, no studies investigated its efficacy in hospitalized patients. Such knowledge will improve patient's compliance and outcomes.

* Sample size calculation: Primary outcome of return to normal activities within 3 days of discharge. Based on previous studies, it is estimated that 70% of the control group will achieve this goal. Based on a minimum absolute difference of 15%, and a power of 0.80, the sample size calculated to be 117 in each arm. Assuming 20% lost to follow up, it is intended to recruit 150 in each arm (total 300 subjects).
* Statistical Analysis: Demographics will be analyzed to ensure the experimental and control groups are equivalent at baseline. All proportions will be tested with Chi-square or Fisher exact test and two-sample T-test will be used for continuous variables. α = 0.05 will be used for all hypothesis tests. Interim analysis will be performed monthly and the study will be halted if any safety concerns arise. The Center for Health Equity and Quality Research (CHEQR) will help with statistical analysis
* Data Safety and Monitoring Plan: The study PI and co-investigator will meet and review the collected data on a monthly basis and identify any interim results that may require a change of study protocol. Information that may affect subjects' safety will be communicated to appropriate parties in a timely fashion.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent by legal guardian
* Age 2 to 18 years old
* Admission to the floor with acute asthma exacerbation.
* Received single dose of oral Dexamethasone
* Initial Pediatric Asthma Score (PAS) of 8 or higher.

Exclusion Criteria:

* Admission to PICU
* Recent steroid use (within 1 month)
* Cardiac disorder, chronic respiratory illness (BPD or CF)
* Stridor
* Bacterial Pneumonia

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2017-08-29 (Actual); Study Completion 2017-08-29 (Actual)

PRIMARY OUTCOMES:
Return to normal activity (Patient Self-Assessment Score) | 3 days after discharge
  Proportion of patients who have returned to normal activity

SECONDARY OUTCOMES:
Relapse ( ED visit or unscheduled physician visit) | 2 weeks after discharge
  Proportion of patients with unscheduled primary care physician visits, emergency department or hospital admission
Albuterol use (Patient Self-Assessment Score) | 2 weeks after discharge
  Proportion of patients with of ongoing albuterol use (based on validated self-reporting tool)
Asthma symptoms (Patient Self-Assessment Score) | 2 weeks after discharge
  Patient self assessment score at 2 weeks after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey C Winer, MD, Principal Investigator — Universiry of Florida, College of Medicine Jacksonville
Locations (1):
- Wolfson Children Hospital, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] National Asthma Education and Prevention Program. Expert Panel Report 3 (EPR-3): Guidelines for the Diagnosis and Management of Asthma-Summary Report 2007. J Allergy Clin Immunol. 2007 Nov;120(5 Suppl):S94-138. doi: 10.1016/j.jaci.2007.09.043. PMID 17983880
- [Background] Keeney GE, Gray MP, Morrison AK, Levas MN, Kessler EA, Hill GD, Gorelick MH, Jackson JL. Dexamethasone for acute asthma exacerbations in children: a meta-analysis. Pediatrics. 2014 Mar;133(3):493-9. doi: 10.1542/peds.2013-2273. Epub 2014 Feb 10. PMID 24515516
- [Background] Qureshi F, Zaritsky A, Poirier MP. Comparative efficacy of oral dexamethasone versus oral prednisone in acute pediatric asthma. J Pediatr. 2001 Jul;139(1):20-6. doi: 10.1067/mpd.2001.115021. PMID 11445789
- [Background] Rowe BH, Spooner CH, Ducharme FM, Bretzlaff JA, Bota GW. Corticosteroids for preventing relapse following acute exacerbations of asthma. Cochrane Database Syst Rev. 2007 Jul 18;2007(3):CD000195. doi: 10.1002/14651858.CD000195.pub2. PMID 17636617
- [Background] Butler K, Cooper WO. Adherence of pediatric asthma patients with oral corticosteroid prescriptions following pediatric emergency department visit or hospitalization. Pediatr Emerg Care. 2004 Nov;20(11):730-5. doi: 10.1097/01.pec.0000144914.78124.6f. PMID 15502653
- [Background] Czock D, Keller F, Rasche FM, Haussler U. Pharmacokinetics and pharmacodynamics of systemically administered glucocorticoids. Clin Pharmacokinet. 2005;44(1):61-98. doi: 10.2165/00003088-200544010-00003. PMID 15634032
- [Background] Gries DM, Moffitt DR, Pulos E, Carter ER. A single dose of intramuscularly administered dexamethasone acetate is as effective as oral prednisone to treat asthma exacerbations in young children. J Pediatr. 2000 Mar;136(3):298-303. doi: 10.1067/mpd.2000.103353. PMID 10700684
- [Background] Klig JE, Hodge D 3rd, Rutherford MW. Symptomatic improvement following emergency department management of asthma: a pilot study of intramuscular dexamethasone versus oral prednisone. J Asthma. 1997;34(5):419-25. doi: 10.3109/02770909709055384. PMID 9350159
- [Background] Gordon S, Tompkins T, Dayan PS. Randomized trial of single-dose intramuscular dexamethasone compared with prednisolone for children with acute asthma. Pediatr Emerg Care. 2007 Aug;23(8):521-7. doi: 10.1097/PEC.0b013e318128f821. PMID 17726409
- [Background] Altamimi S, Robertson G, Jastaniah W, Davey A, Dehghani N, Chen R, Leung K, Colbourne M. Single-dose oral dexamethasone in the emergency management of children with exacerbations of mild to moderate asthma. Pediatr Emerg Care. 2006 Dec;22(12):786-93. doi: 10.1097/01.pec.0000248683.09895.08. PMID 17198210
- [Background] Greenberg RA, Kerby G, Roosevelt GE. A comparison of oral dexamethasone with oral prednisone in pediatric asthma exacerbations treated in the emergency department. Clin Pediatr (Phila). 2008 Oct;47(8):817-23. doi: 10.1177/0009922808316988. Epub 2008 May 8. PMID 18467673
- [Background] National Asthma Education and Prevention Program. National Asthma Education and Prevention Program. Expert Panel Report: Guidelines for the Diagnosis and Management of Asthma Update on Selected Topics--2002. J Allergy Clin Immunol. 2002 Nov;110(5 Suppl):S141-219. No abstract available. PMID 12542074